CLINICAL TRIAL: NCT05264038
Title: A Phase 1, Randomized, Double-Blind, Dose-Ranging, Placebo-controlled Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics Effects of OC514 in Healthy Adult Volunteers
Brief Title: A First in Human Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics Effects of OC514
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncocross Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Organization: Oncocross Co. Ltd. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: OC514-001
Record Dates: First submitted 2022-01-28; First posted 2022-03-03 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Cancer Cachexia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants will receive either low dose level of OC514 or placebo
  Interventions: Drug: OC514 (Low dose); Other: Placebo
- Cohort 2 (Experimental): Participants will receive either mid dose level of OC514 or placebo
  Interventions: Drug: OC514 (Mid dose); Other: Placebo
- Cohort 3 (Experimental): Participants will receive either high dose level of OC514 or placebo
  Interventions: Drug: OC514 (High dose); Other: Placebo

INTERVENTIONS:
Drug: OC514 (Low dose) — Low dose level of OC514
  Other Names: OC514
  Arms: Cohort 1
Drug: OC514 (Mid dose) — Mid dose level of OC514
  Other Names: OC514
  Arms: Cohort 2
Drug: OC514 (High dose) — High dose level of OC514
  Other Names: OC514
  Arms: Cohort 3
Other: Placebo — Placebo to match

SUMMARY:
Oncocross is developing OC514, a drug-drug combination product containing 2 active pharmaceutical ingredients for cancer cachexia. This study is designed to assess the safety and tolerability of single and multiple oral doses of OC514 in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a single-center study in which a total of 24 subjects will be enrolled into 1 of 3 dose level cohorts in an ascending fashion. Each cohort will consist of 8 subjects randomized to receive OC514 or matching placebo at a ratio of 3:1. Eligible subjects will be admitted to the clinical research unit (CRU) from Day -1 to 5 and again from Day 15 to Day 17 and will be discharged upon completion of post-dose assessment. The subjects will attend the CRU for outpatients visits on Day 8 and Day 12. The subjects will return for a follow-up visit on Day 19 and End of Study visit on Day 21.

The total study duration is up to 9 weeks consisting of up to 6 weeks of screening, 2 weeks of blinded treatment, and 1 week of safety follow-up.

Safety oversight will be provided by a Safety Review Committee (SRC).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers, between 18 and 65 years of age, both inclusive.
2. BMI between 18 and 32 kg/m2 (inclusive) with a bodyweight >/= 50 kg at screening.
3. Medically healthy with no clinically significant medical history.
4. Adequate venous access.
5. Non-pregnant, non-lactating females.
6. Must be able to comply with the requirements of the study.

Exclusion Criteria:

1. History of any clinically significant disease or disorder.
2. History or presence of gastrointestinal, hepatic, or renal disease or any other condition or past surgical intervention (eg, cholecystectomy).
3. Has creatinine clearance < 60 mL/min.
4. Any current active infections, including localized infections, or any recent history (within 2 weeks prior to first IP administration) of active infections (including severe acute respiratory syndrome coronavirus 2 [SARS-COV-2]), cough or fever, or a history of recurrent or chronic infections.
5. Lymphoma, leukemia, or any malignancy within the past 5 years except for fully resected basal cell or squamous epithelial carcinomas of the skin that have been fully treated for at least 1 year with no recurrence.
6. Any positive laboratory-confirmed COVID-19 test at Screening or check-in.
7. History of human immunodeficiency virus (HIV) antibody positive or tested positive for HIV; had a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tested positive for HBsAg or anti-HCV at Screening.
8. Had major surgery (general anesthetic) in the last 3 months or minor surgery (local anesthetic) in the last 1 month prior to Screening.
9. History of narrow angle glaucoma.
10. History of benign prostatic hyperplasia (BPH) with lower urinary tract symptoms.
11. Any clinically significant medical or psychiatric condition, medical/surgical procedure, or trauma within 4 weeks prior to the first IP administration.
12. Blood donation within 1 month of Screening or any blood donation/blood loss greater than 500 mL during the 3 months prior to Screening.
13. Abnormal vital signs.
14. Prolonged Fridericia QT correction formula (QTcF) > 450 msec or shortened QTcF < 340 msec or family history of long QT syndrome at the Screening and on Day -1.
15. Positive screen for drugs of abuse or cotinine (≥ 500 ng/mL) or positive screen for alcohol at Screening or admission to the CRU on Day -1.
16. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator, to any components in the IP.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Number of treatment-emergent adverse events (TEAEs) and treatment related TEAEs | Day 1- Day 21
  TEAEs will be measured as per the Common Terminology Criteria for Adverse Events (CTCAE) v 5.0
Severity of TEAEs and treatment related TEAEs | Day 1- Day 21
  TEAEs will be measured as per the Common Terminology Criteria for Adverse Events (CTCAE) v 5.0
Number of participants with abnormal clinically significant laboratory results | Day 1 - Day 21
  Clinical laboratory includes hematology, and biochemistry
Number of patients with abnormal vital signs | Day 1- Day 21
  Includes supine systolic and diastolic blood pressure, pulse rate, oxygen saturation, body temperature, and respiratory rate
Number of participants with abnormal and clinically significant electrocardiogram (ECG) | Day 1 - Day 21
  12-lead ECG will be taken
Number of participants with abnormal urinalysis | Day 1- Day 21
  Dipstick test will be performed
Number of participants with abnormal coagulation test | Day 1- Day 21
  Prothrombin time, International normalization ratio, Activated partial thromboplastin time

SECONDARY OUTCOMES:
Cmax | Day 1-Day 4, Day 8, Day 16, Day 17
  Maximum concentration of OC514 in blood plasma
Tmax | Day 1-Day 4, Day 8, Day 16, Day 17
  Time to maximum concentration
Cmin | Day 1-Day 4, Day 8, Day 16, Day 17
  Minimum concentration
AUC (0-last) | Day 1-Day 4, Day 8, Day 16, Day 17
  Area under the time concentration curve from time zero to last measurable concentration
AUC (0-inf) | Day 1 and Day 2
  AUC from time zero to infinity
AUC (0-12) | Day 3-Day 16
  AUC from time zero until 12 hours post dose
t1/2 | Day 1-Day 4, Day 8, Day 16, Day 17
  Elimination half life
λz or Kel | Day 1-Day 4, Day 8, Day 16, Day 17
  Apparent terminal elimination rate
CL/F and CL/Fss | Day 1-Day 4, Day 8, Day 16, Day 17
  Apparent clearance
Vz/F and Vz/Fss | Day 1-Day 4, Day 8, Day 16, Day 17
  Volume of distribution
Effect of OC514 administration on QT prolongation | Day 4, Day 8, Day 12, Day 16, Day 17, day 19
  12-lead ECG will be done

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Gonen, Dr., Principal Investigator — Nucleus Network
Locations (1):
- Nucleus network, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No